CLINICAL TRIAL: NCT02668640
Title: Real-World Outcome of Adalimumab on Rheumatoid Arthritis Patients in China (ROCKI Study)
Brief Title: Real-World Outcome of Adalimumab on Rheumatoid Arthritis Patients in China
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-776
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Quality of life (QOL); Rheumatoid arthritis (RA); Work productivity; Adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with RA receiving adalimumab: 40 mg adalimumab via subcutaneous (SC) injection every other week (eow) for 24 weeks
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
The objective of this study was to assess the effectiveness of adalimumab on health and disability outcomes in participants with rheumatoid arthritis (RA) in China.

DETAILED DESCRIPTION:
This was a prospective, multicenter, observational study to assess the effectiveness of adalimumab on health-related quality of life (QoL) and work productivity in participants with rheumatoid arthritis (RA) in routine clinical practice in China. The decision to prescribe adalimumab for RA was based on clinical practice criteria without taking participation in this study into account. Participants were included in the study after a physician's decision of initiating adalimumab treatment. Participants were followed for 24 weeks, with scheduled study visits at baseline, Week 12 and Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Participant had a diagnosis of rheumatoid arthritis (RA) as defined by the 1987 revised American College of Rheumatology (ACR) classification criteria and/or the ACR/the European League against Rheumatism (EULAR) 2010 classification criteria (any duration since diagnosis)
* Participants with moderate to severe RA defined as a Disease Activity Score in 28 Joints (DAS28) Erythrocyte Sedimentation Rate (ESR) or DAS28 C-Reactive Protein (CRP) score >3.2
* Biologically treatment naïve and initiated adalimumab at baseline visit, as per standard daily clinical practice
* Availability of clinical data of the previous 12 weeks prior to baseline
* Ability to self-complete participant questionnaires.
* Participants had signed the authorization (or informed consent where applicable) to disclose and use personal health information after having been prescribed adalimumab

Exclusion Criteria:

* Participants who were pregnant or breastfeeding at enrollment or wished to become pregnant in the next 24 weeks.
* Participation in any RA-related clinical trial at the time of enrollment, at baseline, or at any point during the past 24 weeks prior to baseline
* Participants, who in the clinician's view, may not have been able to accurately report their quality of life (QoL) or prior resource utilization
* Participants, who in the clinician's view, may not have been able to adhere to adalimumab therapy over 24 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with rheumatoid arthritis (RA) in China receiving adalimumab treatment
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who received at least one dose of adalimumab during the study
Period: Overall Study
Arm/Group | Participants With RA Receiving Adalimumab
Started | 55
Completed | 41
Not Completed | 14
Not completed — Lost to Follow-up | 13
Not completed — Other, not specified | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of adalimumab during the study
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Medical insurance type [Count of Participants; unit: Participants]
  National/Public insurance | 45
  Private insurance | 2
  Employer benefits | 1
  Other | 5
  No insurance | 1
  National/Public insurance and private insurance | 1
Mean Baseline DAS28 score [Mean (Standard Deviation); unit: units on a scale] — The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) level, and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the score. Scores range from 0 to 10; higher scores indicate more disease activity. A DAS28 score >5.1 indicates high disease activity, a score <3.2 indicates low disease activity, and a score <2.6 indicates clinical remission.
  units on a scale | 6.0 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Median Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) Score at Week 24
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A negative median indicates improvement from baseline.
Time Frame: Baseline and Week 24
Population: Observed population: participants continuing adalimumab treatment after the baseline visit; participants with available data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 39
units on a scale | -0.3 [-0.9 to 0]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Test type: Other; p = 0.0002, Wilcoxon signed-rank test

2. Secondary Outcome: Median Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) Score at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 46
units on a scale | -0.2 [-0.9 to 0]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Test type: Other; p = 0.0006, Wilcoxon signed-rank test

3. Secondary Outcome: Median Change From Baseline in Short Form 36-Item Health Survey (SF-36) Physical Component Summary (PCS) Score and Mental Component Summary (MCS) Scores at Weeks 12 and 24
Description: The SF-36v2 is a non-disease specific Health Related Quality of Life (HRQoL) instrument. The SF-36v2 comprises 36 total items (questions) targeting a subject's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) with a recall period of four weeks. Domain scores are aggregated into a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. SF-36v2 PCS and MCS scores range from 1-100: higher scores indicate a better state of health and an increase from baseline represents improvement.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
units on a scale
  PCS T-Score Week 12: number analyzed (Participants) | 46
  PCS T-Score Week 12 | 6.50 [2.07 to 9.36]
  MCS T-Score Week 12: number analyzed (Participants) | 46
  MCS T-Score Week 12 | 0.44 [-3.49 to 11.00]
  PCS T-Score Week 24: number analyzed (Participants) | 39
  PCS T-Score Week 24 | 4.90 [-2.21 to 11.92]
  MCS T-Score Week 24: number analyzed (Participants) | 39
  MCS T-Score Week 24 | 6.01 [0.00 to 13.35]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Median change from baseline in PCS T-score at Week 12; Test type: Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab; Median change from baseline in MCS T-score at Week 12; Test type: Other; p = 0.1233, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab; Median change from baseline in PCS T-score at Week 24; Test type: Other; p < 0.001, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab; Median change from baseline in MCS T-score at Week 24; Test type: Other; p = 0.001, Wilcoxon signed-rank test

4. Secondary Outcome: Median Change From Baseline in EuroQol 5-dimension, 3-level Quality of Life Questionnaire (EQ-5D-3L) Index
Description: The EQ-5D-3L measures the participant's overall health state in a descriptive system of health-related quality of life (QoL) states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which has three response choices. The responses record three levels of severity ('no problems', 'having some or moderate problems', and 'being unable to do/extreme problems') within a particular EQ-5D-3L dimension. In addition, a 20 cm visual analogue scale (VAS) measures the participant's self-rated current health state on a scale from 0-100, from 0 (worst imaginable health state) to 100 ('best imaginable health state). The EQ-5D-3L results were converted into a weighted health state index with scores ranging from approximately 0 (death) to 1 (full health). A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
units on a scale
  Week 12: number analyzed (Participants) | 46
  Week 12 | 0.11 [0.07 to 0.26]
  Week 24: number analyzed (Participants) | 39
  Week 24 | 0.19 [0.10 to 0.32]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Median Change From Baseline in EQ-5D-3L Index Score at Week 12; Test type: Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab; Median Change From Baseline in EQ-5D-3L Index Score at Week 24; Test type: Other; p < 0.0001, Wilcoxon signed-rank test

5. Secondary Outcome: Median Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Overall Work Impairment Score
Description: The Work Productivity and Activity Impairment Questionnaire (WPAI) is a participant-reported questionnaire to measure work and activity impairment during the past seven days. The 'overall work impairment due to health problem' was calculated based on three items: (Q2) the number of hours missed from work due to health problems in the past seven days from visit; (Q4) the number of actual work hours in the past seven days from visit; and (Q5) to what degree did the participant's rheumatoid arthritis impair the productivity while working past seven days from visit). Data were calculated using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)] and converted to percent, with higher numbers indicating greater impairment and less productivity. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, and Week 24
Population: Observed population: participants continuing adalimumab treatment after the baseline visit who had at least Baseline data for this endpoint
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
percent impairment
  Week 12: number analyzed (Participants) | 10
  Week 12 | -58.4 [-90.0 to -16.7]
  Week 24: number analyzed (Participants) | 9
  Week 24 | -20.0 [-53.3 to 0]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Median Change from Baseline in WPAI Overall Work Impairment Score at Week 12; Test type: Other; p = 0.0137, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab; Median Change from Baseline in Overall Work Impairment Score at Week 24; Test type: Other; p = 0.0607, Wilcoxon signed-rank test

6. Secondary Outcome: Median Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Activity Impairment Score
Description: The Work Productivity and Activity Impairment Questionnaire (WPAI) is a participant-reported questionnaire to measure work and activity impairment during the past seven days. Activity impairment was calculated via WPAI question 6, the participant's rating of how much rheumatoid arthritis affected their ability to do regular daily activities, other than working at a job (0 = no effect; 10 = completely impacted productivity) / 10 * 100. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
percent impairment
  Week 12: number analyzed (Participants) | 45
  Week 12 | -10.0 [-30.0 to -10.0]
  Week 24: number analyzed (Participants) | 38
  Week 24 | -20.0 [-30.0 to 0.0]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab; Median Change from Baseline in WPAI Activity Impairment Score at Week 12; Test type: Other; p = 0.0026, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab; Median Change from Baseline in WPAI Activity Impairment Score at Week 24; Test type: Other; p = 0.0001, Wilcoxon signed-rank test

7. Secondary Outcome: Number of Participants Achieving Clinically Meaningful Improvement in Health Assessment Questionnaire- Disability Index (HAQ-DI) Score
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥ 0.22.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
Participants
  Week 12: number analyzed (Participants) | 46
  Week 12 | 23
  Week 24: number analyzed (Participants) | 39
  Week 24 | 20

8. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Improvement in Health Assessment Questionnaire- Disability Index (HAQ-DI) Score
Description: as for outcome 7
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 54
percentage of participants
  Week 12: number analyzed (Participants) | 46
  Week 12 | 50.0
  Week 24: number analyzed (Participants) | 39
  Week 24 | 51.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 70 days after the last dose of study drug (up to 34 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of adalimumab is administered until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Participants With RA Receiving Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 2/55
Other Adverse Events (participants affected / at risk) | 17/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With RA Receiving Adalimumab (N=55)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With RA Receiving Adalimumab (N=55)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Injection site hypersensitivity (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT02668640/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02668640/SAP_001.pdf